CLINICAL TRIAL: NCT03217435
Title: A Non-randomized Controlled Clinical Trial of Epithelial Allograft Transplantation From Living-related Donors for the Treatment of Limbal Stem Cell Deficiency
Brief Title: Corneal Epithelial Allograft From Living-related Donor for LSCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chunxiao Wang (Other)
Responsible Party: Sponsor-Investigator, Chunxiao Wang, Clinical investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017KYPJ057
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cornea epithelial allograft (Experimental): Femtosecond laser assisted corneal epithelial allograft from live relatives in the treatment of limbal stem cell deficiency (LSCD)
  Interventions: Procedure: Corneal epithelial allograft; Device: Femtosecond laser
- Limbal conjunctival allograft (Active Comparator): Diamond knife assisted limbus conjunctival allograft from live relatives in the treatment of limbal stem cell deficiency (LSCD)
  Interventions: Procedure: Limbal conjunctival allograft; Device: Diamond knife

INTERVENTIONS:
Procedure: Corneal epithelial allograft — A living-related donor's epithelial flap, equal in area to the recipient's diseased cornea bed, will be created using femtosecond laser technology. This corneal epithelial allograft is then ready for transplantation on the recipient's disease eye, following removal of the recipient's scarred and diseased epithelium.
  Arms: Cornea epithelial allograft
Procedure: Limbal conjunctival allograft — A 3- to 5- clock hour limbal-conjunctival allograft will be obtained from the living-related eye. This is then ready for transplantation on the recipient's disease eye following removal of the recipient's scarred and diseased epithelium.
  Arms: Limbal conjunctival allograft
Device: Femtosecond laser — A commercial femtosecond laser to create a particular shaped graft for transplantation
  Arms: Cornea epithelial allograft
Device: Diamond knife — A diamond knife to create a particular shaped limbal graft for transplantation
  Arms: Limbal conjunctival allograft

SUMMARY:
The purpose of the study is to explore whether femtosecond laser-assisted corneal epithelial allograft from living-related donor is more effective than limbal conjunctival allograft from living-related donor for ocular surface reconstruction in patients with limbal stem cell deficiency (LSCD).

ELIGIBILITY:
Inclusion Criteria:

1. LSCD secondary to ocular burns, with the duration of disease of at least 24 months at the time of screening visit;
2. Presence of superficial neo-vascularization affecting at least 2 cornea quadrants and involving central cornea;
3. Having a human leukocyte antigen (HLA)-matched living-related donor (≥4/6 HLA-A/B/DR matched);
4. Informed consent signed by patient or legal guardian. Having the ability to comply with study assessments for the full duration of the study.

Exclusion Criteria:

Recipients:

1. LSCD of mild degree, with less than 2 quadrants of neo-vessel invasion and without central cornea involvement;
2. LSCD by ocular surface disorders other than ocular burn;
3. Eyelids malposition;
4. The center corneal thickness<450µm, the depth of corneal opacity > 150µm;
5. High myopia with a spherical equivalent of -15.0 D or less;
6. Corneal or ocular surface infection within 30 days prior to study entry;
7. Ocular surface malignancy;
8. Uncontrolled diabetes with most recent Hemoglobin A1c greater than 8.5%;
9. Renal failure with creatinine clearance< 25ml/min;
10. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L;
11. Platelet levels < 150,000 or > 450,000 per microliter;
12. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female);
13. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy; An international normalized ratio greater than 3 in patients accepting anticoagulant therapy;
14. Pregnancy (positive test) or lactation;
15. Participation in another simultaneous medical investigation or clinical trial;
16. Severe cicatricial eye disease; Conjunctival scarring with fornix shortening;
17. Ocular comorbidities that affect the prognosis of transplantation, such as advanced glaucoma or retinal diseases;
18. Severe dry eye disease as determined by Schirmer's test < 2mm at least in one eye;
19. Any medical or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent;
20. Signs of current infection, including fever and treatment with antibiotics;
21. Active immunological diseases;
22. History of allo-limbal transplantation, penetrating keratoplasty or anti-glaucoma filtering surgeries.

Donors:

1. Cornea diseases (epithelial defects, neovascularization, etc.);
2. Eyelids malposition;
3. The center corneal thickness<450µm, the depth of corneal opacity > 150µm;
4. High myopia with a spherical equivalent of -15.0 D or less;
5. Corneal or ocular surface infection within 30 days prior to study entry;
6. Ocular surface malignancy;
7. Uncontrolled diabetes with most recent Hemoglobin A1c greater than 8.5%;
8. Renal failure with creatinine clearance< 25ml/min;
9. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L;
10. Platelet levels < 150,000 or > 450,000 per microliter;
11. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female);
12. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy; An international normalized ratio greater than 3 in patients accepting anticoagulant therapy;
13. Pregnancy (positive test) or lactation;
14. Participation in another simultaneous medical investigation or clinical trial;
15. Severe cicatricial eye disease; Conjunctival scarring with fornix shortening;
16. Ocular comorbidities that affect the prognosis of transplantation, such as advanced glaucoma or retinal diseases;
17. Severe dry eye disease as determined by Schirmer's test < 2mm at least in one eye;
18. Any medical or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent;
19. Signs of current infection, including fever and treatment with antibiotics;
20. Active immunological diseases;
21. History of allo-limbal transplantation, penetrating keratoplasty or anti-glaucoma filtering surgeries.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Restoration of corneal surface in the recipient | 1 year
  Restoration of a completely epithelized, stable, and avascular corneal surface in the recipient
Restoration of corneal surface in the donor | 1 year
  Restoration of a completely epithelized, stable, and avascular corneal surface in the donor

SECONDARY OUTCOMES:
Uncorrected and best-corrected visual acuity of recipients and donors | 1 year
  To assess changes of uncorrected and best-corrected visual acuity using ETDRS chart.
Corneal power, astigmatism and aberration of recipients and donors | 1 year
  To measure changes of corneal power, astigmatism and aberration using autorefractor keratometer and wavefront aberrometer respectively.
Corneal sensation of recipients and donors | 1 year
  To measure corneal sensation using Cochet-Bonnet esthesiometer.
Corneal thickness of recipients and donors | 1 year
  To measure corneal thickness using Anterior Segment Optical Coherence Tomograph (AS-OCT).
Density of stromal nerve and stromal keratocytes of recipients and donors | 1 year
  To measure density of stromal nerve and stromal keratocytes using in vivo confocal microscopy
Reconstruction of limbal palisades of Vogt of recipients | 1 year
  To assess reconstruction of limbal palisades of Vogt using in vivo confocal microscopy.
Corneal graft rejection of recipients | 1 year
  To assess corneal graft rejection using slit-lamp microscopy.
Corneal haze of recipients and donors | 1 year
  To assessing corneal haze using in vivo confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Ting Huang, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China